CLINICAL TRIAL: NCT04073550
Title: A Randomized, Double-Blind, Multicenter, Phase Ⅲ Study of Anlotinib Hydrochloride Capsule Combined With Topotecan Versus Placebo Combined With Topotecan in Subjects With Small Cell Lung Cancer
Brief Title: Study of Anlotinib Hydrochloride Capsule in Subjects With Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-12-III-01
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib; Topotecan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Anlotinib hydrochloride capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) and topotecan 1.5mg/m2 IV d1-5.
  Interventions: Drug: Anlotinib; Drug: Topotecan
- Placebo group (Placebo Comparator): Anlotinib hydrochloride placebo given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) and topotecan 1.5mg/m2 IV d1-5.
  Interventions: Drug: Placebos; Drug: Topotecan

INTERVENTIONS:
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor.
  Arms: Experimental group
Drug: Placebos — Anlotinib blank analog capsule.
  Arms: Placebo group
Drug: Topotecan — A topoisomerase I inhibitor.

SUMMARY:
Anlotinib hydrochloride is a multi-targeted receptor tyrosine kinase inhibitor that targets angiogenesis-related kinases such as VEGFR1/2/3, FGFR1/2/3, and other tumor-associated kinases involved in cell proliferation such as PDGFRα/β, c-Kit, and Ret have significant inhibitory activities.

ELIGIBILITY:
Inclusion Criteria:

1. Small cell lung cancer patients.
2. The clinical stage at baseline is extensive.
3. A measurable lesion.
4. Disease progression.
5. ≥ 18 years old; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.
6. Adequate laboratory indicators.
7. No pregnant or breastfeeding women, and a negative pregnancy test.
8. Understood and signed an informed consent form.

Exclusion Criteria:

1. Has used topotecan and anlotinib hydrochloride capsules.
2. Has used other anti-angiogenic drugs and immunologically targeted drugs.
3. Has other malignant tumors within 5 years.
4. Symptomatic brain metastasis.
5. Has a variety of factors affecting oral medications.
6. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage.
7. Spinal cord compression.
8. Has received radiotherapy, chemotherapy, surgery less than 4 weeks before randomization.
9. Adverse events caused by previous treatment did not recover to grade 1.
10. Has received major surgical treatment within 4 weeks before randomization.
11. Arteriovenous thrombosis occurred within 6 months.
12. Has drug abuse history that unable to abstain from or mental disorders.
13. Has severe or uncontrolled disease.
14. Participated in other clinical trials within 4 weeks.
15. Tumor invades the large blood vessels.
16. Daily hemoptysis ≥2.5 mL within 1 month before the first dose.
17. According to the investigators' judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-10-31 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) evaluated by IRC | up to 24 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause; IRC defined as Independent Review Committee.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) evaluated by investigator | up to 24 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to 24 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Overall Response Rate (ORR) | up to 24 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR).
Disease Control Rate (DCR) | up to 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Overall Response (DOR) | up to 24 months
  The time when the patient first achieved complete or partial remission to disease progression.
PFS rate at month 6 | up to 6 months
  The percentage of PFS at month 6.
OS rate at month 6 | up to 6 months
  The percentage of OS at month 6.
OS rate at month 12 | up to 12 months
  The percentage of OS at month 12.
The efficacy of intracranial lesions | up to 24 months
  To evaluate the efficacy of of intracranial lesions.
Adverse Event (AE) | up to 24 months
  Safety data
Serious Adverse Event (SAE) | up to 24 months
  Safety data
Abnormal laboratory test index | up to 24 months
  Safety data

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality